CLINICAL TRIAL: NCT01198873
Title: A Placebo-Controlled, Double-Blind, Randomized, Multi-center Study to Assess the Effects of Dronedarone 400 mg BID on Cardiac Geometry and Function in Patients With Atrial Fibrillation and Left Atrial Enlargement
Brief Title: Effects of Dronedarone on Cardiac Geometry and Function in Patients With Atrial Fibrillation and Left Atrial Enlargement
Acronym: ODYSSEUS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DRONE_L_04315
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Results first posted 2013-02-12 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dronedarone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dronedarone (Experimental): Dronedarone 400 mg twice a day
  Interventions: Drug: Dronedarone
- Placebo (Placebo Comparator): Placebo (for Dronedarone) twice a day
  Interventions: Drug: Placebo (for Dronedarone)

INTERVENTIONS:
Drug: Dronedarone — Film-coated tablet
  Oral administration under fed conditions (during breakfast and dinner)
  Other Names: Multaq®; SR33589
  Arms: Dronedarone
Drug: Placebo (for Dronedarone) — film-coated tablet strictly identical in appearance
  Oral administration under fed conditions (during breakfast and dinner)
  Arms: Placebo

SUMMARY:
Primary Objective:

- Evaluate the effect of dronedarone versus placebo (standard therapy) in slowing the progression of adverse left atrial remodeling in patients with atrial fibrillation (AF) following 12 months of treatment.

Secondary Objectives:

* Evaluate the effects of dronedarone versus placebo on left atrial function;
* Evaluate the effects of dronedarone versus placebo on left atrial dimension;
* Evaluate the effects of dronedarone versus placebo on left ventricular function (LVEF, E, E', A, E/E')
* Evaluate the safety and tolerability of dronedarone.

DETAILED DESCRIPTION:
The planned total study period per participant was 12 months and 3 weeks broken down as follows:

* Screening period: up to 1 week;
* Treatment period: 12 months;
* Follow-up period: 2 weeks.

ELIGIBILITY:
Inclusion criteria:

* Signed written informed consent and Health Insurance Portability and Accountability Act (HIPAA) Authorization;
* Nonpermanent AF or AF/Atrial Flutter (AFL) documented electrocardiographically by both AF (or AF/AFL) and sinus rhythm within the prior 12 months;
* At screening, sinus rhythm and Left Atrial Volume index (LAVi) ≥32 mL/m2 based on 2D-echocardiography;
* At least one of the following cardiovascular (CV) risk factors: Age >70 years at start of screening, hypertension, diabetes mellitus, prior CV accident (stroke or transient ischemic attack) or systemic embolism, or left ventricular ejection fraction <0.40.

Exclusion criteria:

* Permanent AF defined as continuous AF for 6 months or longer;
* Persistent AF defined as sustained AF >7 days duration and/or requiring cardioversion in the 4 weeks before screening;
* Prior valvular heart surgery or significant valvular heart disease including rheumatic heart disease or acquired valvular heart disease;
* Aortic or mitral regurgitation greater than mild (>1+) or any degree of mitral stenosis at the screening echocardiogram;
* Myocardial infarction within the 6 months prior to screening or stroke within 2 months prior to screening;
* Pacemaker, implantable cardioverter defibrillator, or cardiac resynchronization therapy devices placed within the 6 months prior to screening or at anytime during the study;
* Ongoing potentially dangerous symptoms when in AF/AFL such as angina pectoris, transient ischemic attacks, stroke, syncope as judged by the Investigator;
* Cardiac ablative procedure or cardiac surgery within 3 months prior to screening, or percutaneous coronary intervention within 4 weeks prior to screening;
* Need for concomitant medication that is prohibited in this trial, and would preclude the use of the study drug during the planned study period including the following:

  * Antiarrhythmics (eg, amiodarone, flecainide, propafenone, quinidine, disopyramide, dofetilide, sotalol);
  * Drugs or products that are strong inhibitors of CYP3A (eg, ketoconazole, itraconazole, voriconazole, cyclosporine, telithromycin, clarithromycin, nefazodone, ritonavir, and grapefruit juice);
  * Drugs that are inducers of CYP3A (eg, rifampin, phenobarbital, carbamazepine, phenytoin, and St John's wort);
* QTc Bazett interval ≥500 msec on the screening ECG;
* Bradycardia <50 bpm and/or PR interval ≥0.28 sec on the screening ECG unless the patient has a functional pacemaker;
* New York Heart Association (NYHA) Class IV heart failure or NYHA Class II or III heart failure with a recent decompensation requiring hospitalization or referral to a specialized heart failure clinic within 4 weeks prior to screening.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2010-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (57):
- United States (56):
  - Investigational Site Number 840072, Phoenix, Arizona
  - Investigational Site Number 840015, Little Rock, Arkansas
  - Investigational Site Number 840086, Beverly Hills, California
  - Investigational Site Number 840018, Loma Linda, California
  - Investigational Site Number 840029, Merced, California
  - Investigational Site Number 840044, Redwood City, California
  - Investigational Site Number 840042, Santa Ana, California
  - Investigational Site Number 840060, Vista, California
  - Investigational Site Number 840057, Stamford, Connecticut
  - Investigational Site Number 840002, Newark, Delaware
  - Investigational Site Number 840063, Wilmington, Delaware
  - Investigational Site Number 840070, Bradenton, Florida
  - Investigational Site Number 840010, Jacksonville, Florida
  - Investigational Site Number 840071, Jupiter, Florida
  - Investigational Site Number 840061, Lakeland, Florida
  - Investigational Site Number 840096, Lauderdale Lakes, Florida
  - Investigational Site Number 840031, Ocala, Florida
  - Investigational Site Number 840074, Orlando, Florida
  - Investigational Site Number 840016, Ormond Beach, Florida
  - Investigational Site Number 840051, St. Petersburg, Florida
  - Investigational Site Number 840081, Roswell, Georgia
  - Investigational Site Number 840103, Jerseyville, Illinois
  - Investigational Site Number 840106, Peoria, Illinois
  - Investigational Site Number 840066, Elkhart, Indiana
  - Investigational Site Number 840099, Lexington, Kentucky
  - Investigational Site Number 840039, Owensboro, Kentucky
  - Investigational Site Number 840092, Baton Rouge, Louisiana
  - Investigational Site Number 840040, Auburn, Maine
  - Investigational Site Number 840077, Ayer, Massachusetts
  - Investigational Site Number 840050, Alpena, Michigan
  - Investigational Site Number 840041, Saginaw, Michigan
  - Investigational Site Number 840058, Minneapolis, Minnesota
  - Investigational Site Number 840101, Picayune, Mississippi
  - Investigational Site Number 840078, St Louis, Missouri
  - Investigational Site Number 840038, St Louis, Missouri
  - Investigational Site Number 840102, St Louis, Missouri
  - Investigational Site Number 840012, Kalispell, Montana
  - Investigational Site Number 840090, Lincoln, Nebraska
  - Investigational Site Number 840045, Buffalo, New York
  - Investigational Site Number 840055, Manhasset, New York
  - Investigational Site Number 840003, The Bronx, New York
  - Investigational Site Number 840004, Troy, New York
  - Investigational Site Number 840009, Maumee, Ohio
  - Investigational Site Number 840028, Camp Hill, Pennsylvania
  - Investigational Site Number 840067, Wyomissing, Pennsylvania
  - Investigational Site Number 840027, Wakefield, Rhode Island
  - Investigational Site Number 840046, Knoxville, Tennessee
  - Investigational Site Number 840014, Longview, Texas
  - Investigational Site Number 840068, Danville, Virginia
  - Investigational Site Number 840069, Manassas, Virginia
  - Investigational Site Number 840087, Richmond, Virginia
  - Investigational Site Number 840085, Winchester, Virginia
  - Investigational Site Number 840013, Burien, Washington
  - Investigational Site Number 840091, Spokane, Washington
  - Investigational Site Number 840080, Madison, Wisconsin
  - Investigational Site Number 840023, Milwaukee, Wisconsin
- Investigational Site Number 124003, Cambridge, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment initiated in September 2010 was discontinued in September, 2011 due to significantly lower than planned enrollment with no feasibility to complete the trial within reasonable, meaningful timelines.
  At that time 57 sites in US and Canada had screened at least one patient.
Pre-assignment Details: After signature of the informed consent and after eligibility was confirmed, group assignment was made at site in a 1:1 ratio using a treatment code list generated centrally by Sanofi. Participants were considered as randomized as soon as the assignment was made.
  A total of 76 participants were randomized at 39 sites.
Groups:
- Placebo: Placebo (for Dronedarone) twice a day (average treatment duration of approximatively 6 months)
- Dronedarone: Dronedarone 400 mg twice a day (average treatment duration of approximatively 6 months)
Period: Overall Study
Arm/Group | Placebo | Dronedarone
Started | 41 | 35
Treated | 41 | 35
Evaluable for Efficacy | 33 (8 participants discontinued before completing 3-month treatment and were not assessed post-baseline) | 26 (9 participants discontinued before completing 3-month treatment and were not assessed post-baseline)
Completed | 4 | 3
Not Completed | 37 | 32
Not completed — Adverse Event | 4 | 7
Not completed — Study closure | 29 | 23
Not completed — Other than above | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dronedarone | Total
Number analyzed (Participants) | 41 | 35 | 76
Age Continuous [Mean (Standard Deviation); unit: years] | 70.3 (8.2) | 74.1 (9.7) | 72.0 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 26 | 22 | 48

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Left Atrial Volume Index (LAVi)
Description: Left Atrial Volume index (LAVi) was assessed at baseline and after 12 months treatment using 2-D echocardiography and interpreted blindly via a central Echocardiography Core Lab.
  Participants who discontinued after completing at least 3 months of treatment were assessed after last study drug intake and data were included in the analysis.
Time Frame: baseline (before randomization) and post-baseline (after 3-12 months of treatment)
Population: The analysis included all randomized and treated participants with at least one post-baseline echocardiographic assessment. Participants were included in the treatment group to which they were randomized (Modified Intent-to-treat analysis).
  The quality of the post-baseline echocardiography was inadequate for determining LAVi in one participant.
Measure: Mean (Standard Deviation); unit: mililiters/m2
Arm/Group | Placebo | Dronedarone
Number analyzed (Participants) | 33 | 26
mililiters/m2
  Baseline (n =33, 26) | 37.555 (5.899) | 37.715 (6.597)
  Post-baseline (n =32, 26) | 29.191 (5.994) | 30.823 (5.364)
  Change from baseline (n =32, 26) | -8.438 (4.743) | -6.892 (5.759)

2. Secondary Outcome: Changes From Baseline in Left Atrial Function
Description: left atrial (LA) function was assessed at baseline and after 12 months treatment using 2-D echocardiography and interpreted blindly via a central Echocardiography Core Lab.
  Participants who discontinued after completing at least 3 months of treatment were assessed after last study drug intake and data were included in the analysis.
Time Frame: baseline (before randomization) and post-baseline (after 3-12 months of treatment)
Population: Modified intent-to-treat population as previously defined
Measure: Mean (Standard Deviation); unit: mililiters
Arm/Group | Placebo | Dronedarone
Number analyzed (Participants) | 33 | 26
mililiters
  LA passive emptying volume (n = 19, 19) | -10.783 (7.798) | -4.566 (9.094)
  LA conduit volume (n =29, 25) | -1.366 (5.652) | -0.764 (5.759)
  LA active emptying volume (n = 19, 19) | -0.052 (4.707) | 1.198 (5.695)
  LA passive emptying fraction (n = 19, 19) | -0.074 (0.074) | -0.019 (0.117)
  LA active emptying fraction (n = 19, 19) | 0.057 (0.104) | 0.067 (0.105)

3. Secondary Outcome: Changes From Baseline in Left Atrial Dimension
Description: Maximal left atrial diameter in the anteroposterior dimension was assessed at baseline and after 12 months treatment using 2-D echocardiography and interpreted blindly via a central Echocardiography Core Lab.
  Participants who discontinued after completing at least 3 months of treatment were assessed after last drug intake and data were included in the analysis.
Time Frame: baseline (before randomization) and post-baseline (after 3-12 months of treatment)
Population: Modified intent-to-treat population as previously defined
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Placebo | Dronedarone
Number analyzed (Participants) | 33 | 26
centimeters | -0.124 (0.188) | -0.166 (0.161)

4. Secondary Outcome: Changes From Baseline in Left Ventricular Ejection Fraction (LVEF)
Description: Left Ventricular Ejection Fraction (LVEF) was assessed at baseline and after 12 months treatment using 2-D echocardiography and interpreted blindly via a central Echocardiography Core Lab.
  Participants who discontinued after completing at least 3 months of treatment were assessed after last drug intake and data were included in the analysis.
Time Frame: baseline (before randomization) and post-baseline (after 3-12 months of treatment)
Population: Modified intent-to-treat population as previously defined
Measure: Mean (Standard Deviation); unit: percentage of blood pumped out
Arm/Group | Placebo | Dronedarone
Number analyzed (Participants) | 33 | 26
percentage of blood pumped out | 0.948 (3.333) | 1.147 (3.997)

5. Secondary Outcome: Changes From Baseline in Left Ventricular Function
Description: left ventricular (LV) function was assessed at baseline and after 12 months treatment using 2-D echocardiography and interpreted blindly via a central Echocardiography Core Lab.
  Participants who discontinued after completing at least 3 months of treatment were assessed after last study drug intake and data were included in the analysis.
Time Frame: baseline (before randomization) and post-baseline (after 3-12 months of treatment)
Measure: Mean (Standard Deviation); unit: centimeters/second
Arm/Group | Placebo | Dronedarone
Number analyzed (Participants) | 33 | 26
centimeters/second
  Peak early diastolic transmitral flow velocity (E) | 5.165 (15.440) | -10.497 (27.890)
  Mitral annular velocity (E') | 0.847 (2.002) | -0.119 (1.845)
  Peak late diastolic transmitral flow velocity (A) | 0.076 (11.674) | 4.319 (14.275)
  E/E' ratio | -0.787 (3.346) | -1.443 (4.288)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected regardless of seriousness or relationship to the drug in the period spanning from signature of the Informed Consent Form up to the last visit.
Description: The analysis included all randomized participants who received at least one dose of study drug and all AE that developed or worsened from randomization up to 10 days after last study drug intake.
  Participants were considered according to the treatment actually received regardless the amount of treatment administered.
Arm/Group | Placebo | Dronedarone
Serious Adverse Events (participants affected / at risk) | 1/41 | 5/35
Other Adverse Events (participants affected / at risk) | 5/41 | 14/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | Dronedarone (N=35)
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatic cyst (Gastrointestinal disorders) | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | Dronedarone (N=35)
Pneumonia (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 3
Depression (Psychiatric disorders) | 0 | 2
Dizziness (Nervous system disorders) | 0 | 3
Hypertension (Vascular disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 4
Nausea (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 2
Fatigue (General disorders) | 1 | 4
Oedema peripheral (General disorders) | 2 | 2

LIMITATIONS AND CAVEATS:
Due to the early termination of the study, results should be cautiously interpreted. Indeed the number of participants was lower than planned (76 instead of 334) and the treatment period was shorter than planned (6 months instead of 12 months).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months after trial completion, the Investigator can present or publish trial results. A copy is submitted to the Sponsor for review and comment at least 30 days in advance of any presentation or submission for publication.

The Sponsor can require to delay the communication for a period not exceeding 90 days to allow for filing a patent application or such other measures as Sponsor deems appropriate to establish and preserve its proprietary rights.